CLINICAL TRIAL: NCT05175131
Title: Multicenter, Randomized, Parallel-group, Open-label, Comparative Clinical Study to Evaluate Efficacy and Safety of Mebeverine+Simethicone Fixed-dose Combination Versus Duspatalin® (Mebeverine) and Versus Espumisan® (Simethicone) in Patients With Functional Bowel Disorders With Abdominal Pain and Excess Gas Formation
Brief Title: Efficacy and Safety of Mebeverine + Simethicone in Patients With Functional Bowel Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MESI3001
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Functional Bowel Disorder
Keywords: Mebeverine+Simethicone; Duspatalin; abdominal pain; bloating/flatulence; functional bowel disorder; fixed dose combination; NRS11
MeSH Terms: conditions — Abdominal Pain; Flatulence | interventions — mebeverine; Simethicone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mebeverine+Simethicone combination (Experimental): three times a day per os
  Interventions: Drug: Mebeverine+Simethicone
- mebeverine (Active Comparator): three times a day per os
  Interventions: Drug: Mebeverine
- simethicone (Active Comparator): 80 mg (2 capsules 40 mg) three times a day per os
  Interventions: Drug: Simethicone

INTERVENTIONS:
Drug: Mebeverine+Simethicone — fixed-dose combination, film-coated tablets, 135 mg + 80 mg
  Arms: Mebeverine+Simethicone combination
Drug: Mebeverine — Duspatalin®, coated tablets 135 mg
  Arms: mebeverine
Drug: Simethicone — Espumisan® capsules 40 mg
  Arms: simethicone

SUMMARY:
The parallel three-group study of efficacy and safety was planned to investigate the reduction in abdominal pain and bloating during treatment with the fixed-dose combination of Mebeverine + Simethicone versus Duspatalin® and Espumisan® as a monotherapy (Protocol No. MESI3001).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form;
2. Males and females aged 18 to 75 years old (inclusive);
3. Abdominal pain and bloating/flatulence due to functional bowel disorder (including IBS, chronic functional constipation, chronic functional diarrhea or functional abdominal bloating);
4. Episodes of abdominal pain for at least 3 months, with a frequency of at least 3 times a month;
5. Abdominal pain intensity of 4 to 9 points (inclusive) when assessed on the NRS-11 scale (i.e. weekly average, with daily recording of the worst pain for the last 24 hours during last week of Screening and Run-in period);
6. Bloating/flatulence intensity of of 4 to 9 points (inclusive) when assessed on the NRS-11 scale (i.e. weekly average, with daily recording of the worst bloating episode for the last 24 hours during last week of Screening and Run-in period);
7. Patients' consent to use adequate contraception methods throughout the study. Adequate contraception methods include:

   1. oral contraceptives or contraceptive patches,
   2. condom or diaphragm (barrier method) with spermicide, or
   3. an intrauterine device

Exclusion Criteria:

1. Hypersensitivity to mebeverine, simethicone, drotaverine, excipients of the studied products, or contraindications;
2. Intake of tricyclic antidepressants, eluxadoline, linaclotide, selective serotonin re-uptake inhibitors, rifaximin, lubriprostone within the last week before screening;
3. New prescription or any change in probiotic drug therapy (including change in the drug or dosage regimen) during the last month before screening;
4. History of intestinal obstruction, stricture, toxic megacolon, GI (gastro-intestinal) perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation (e.g. aorto-iliac disease);
5. History of major gastric, hepatic, pancreatic or intestinal surgery (appendectomy, hemorrhoidectomy, or polypectomy allowed as long as occurred > 3 months prior to trial screening; uncomplicated laparoscopic or open cholecystectomy is allowed if no history of post-operative biliary tract pain and surgery occurred > 3 months prior to screening);
6. Significant and progressive enlargement of the liver, spleen, lymph nodes; ascites; palpable tumor formation in the abdominal cavity / pelvis according to physical examination, hepatic cirrhosis;
7. Significant concomitant acute or chronic disease (cardiovascular, gastrointestinal, endocrine, immunological, metabolic, bronchopulmonary, urinary system) or any condition that, according to Investigator, is a contraindication for the patient to participate in the study if interference with the study performance;
8. Any inflammatory bowel disease (Crohn's disease, ulcerative colitis, any infection including bacterial, viral, protozoa, helminthosis);
9. Elevated fecal calprotectin level 1 month before or at screening which indicates the presence of inflammatory GIT disease;
10. Unexplained GI bleeding within 3 months prior to screening;
11. Confirmed diagnosis of bile acids malabsorption;
12. History of any malignant disease except basal cell carcinoma of skin and vesical cervix carcinoma in situ which were cured ≥ 5 years ago;
13. Confirmed diagnosis of celiac disease;
14. Confirmed hereditary galactose or fructose intolerance , total lactase deficiency, sucrase-isomaltose insufficiency, glucose-galactose malabsorption syndrome;
15. Diet changes (e.g, switching to fermented foods, a gluten-free diet) within the 1 months prior to screening;
16. Planned elective surgery during the study;
17. Pancreatic exocrine insufficiency or acute pancreatitis;
18. Endometriosis in women;
19. Positive results of tests for HIV, hepatitis B or C, at the moment of screening;
20. Drugs or alcohol abuse at screening or in the past, which, in the Investigator's opinion, makes the patient not eligible for participation in the study;
21. Participation in another clinical study or another study drug administration within 30 days prior to screening;
22. Pregnant or lactating women, or women planning to get pregnant during the clinical study; women of child-bearing potential (including those without history of surgical sterilization and women with <2 years post-menopause) not using adequate contraception methods;
23. Inability to read or right; unwillingness to understand and comply with Protocol procedures; non-compliance with medication dosing regimen or procedures which, in the Investigator's opinion, may affect study results or the patient's safety and prevent the patient's participation in the study; any other concomitant diseases or severe mental disorders, which make the patient ineligible for study participation, limit the legal basis for Informed Consent procedure, or may affect the patient's ability to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Null Research Facilities, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mebeverine+Simethicone Combination | Mebeverine | Simethicone
Started | 155 | 155 | 155
Completed | 153 | 154 | 152
Not Completed | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mebeverine+Simethicone Combination | Mebeverine | Simethicone | Total
Number analyzed (Participants) | 155 | 155 | 155 | 465
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 151 | 152 | 146 | 449
  >=65 years | 4 | 3 | 9 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 110 | 102 | 315
  Male | 52 | 45 | 53 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 152 | 154 | 154 | 460
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 155 | 155 | 155 | 465

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Sum of NRS-11 Abdominal Pain and Bloating/Flatulence Intensity Scores After 4 Weeks of Treatment.
Description: The baseline abdominal pain and bloating/flatulence intensity was determined as the average of the Numeric rating scale (NRS-11) daily assessment during 7 days before randomization.
  The Week 4 assessment was the average from last 7 days of the corresponding week.
  The scale is a horizontal 10 cm line with the numbers from 0 to 10 located on it, where 0 is "no pain/bloating", 10 is "most severe pain/bloating you can imagine".
Time Frame: 4 weeks
Population: 465 subjects were allocated to treatment. 2 subjects had only a baseline assessment of the efficacy parameters and were excluded from the full analysis sample. Therefore, 463 subjects were included in the Full Analysis Sample (FAS)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mebeverine+Simethicone Combination | Mebeverine | Simethicone
Number analyzed (Participants) | 154 | 155 | 154
score on a scale | -7.23 (3.42) | -6.48 (3.48) | -5.86 (3.72)
Statistical Analysis 1: Comparison: Mebeverine+Simethicone Combination vs Mebeverine; ANCOVA was used for primary end point analysis. The model included the change from baseline of the NRS_11 score as dependent variable and treatment and site as independent factors, and baseline NRS-11 as covariate; Test type: Superiority; p = 0.0042, ANCOVA; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [0.3 to 1.8] — Mean difference of Mebeverine+Simethicone combination to Mebeverine. Adjusted least squares mean (difference between Mebeverine+Simethicone combination and Mebeverine) from ANCOVA is presented here
Statistical Analysis 2: Comparison: Mebeverine+Simethicone Combination vs Simethicone; Mean difference of Mebeverine+Simethicone combination to Simethicone. ANCOVA was used for primary end point analysis. The model included the change from baseline of the NRS_11 score as dependent variable and treatment and site as independent factors, and baseline NRS-11 as covariate; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [0.9 to 2.4] — Adjusted least squares mean (difference between Mebeverine+Simethicone combination and Mebeverine) from ANCOVA is presented here

2. Secondary Outcome: Change From Baseline of NRS-11 Pain Intensity After 4 Weeks of Treatment
Description: The baseline pain intensity was determined as the average of the Numeric rating scale (NRS-11) daily assessment during 7 days before randomization. The Week 4 assessment was the average from last 7 days of the corresponding week.
  The scale is a horizontal 10 cm line with the numbers from 0 to 10 located on it, where 0 is "no pain/bloating", 10 is "most severe pain/bloating you can imagine".
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mebeverine+Simethicone Combination | Mebeverine | Simethicone
Number analyzed (Participants) | 154 | 155 | 154
score on a scale | -3.59 (1.77) | -3.19 (1.80) | -2.75 (1.88)

3. Secondary Outcome: Change From Baseline of NRS-11 Bloating/Flatulence Intensity After 4 Weeks of Treatment
Description: The baseline bloating/flatulence intensity was determined as the average of the Numeric rating scale (NRS-11) daily assessment during 7 days before randomization. The Week 4 assessment was the average from last 7 days of the corresponding week.
  The scale is a horizontal 10 cm line with the numbers from 0 to 10 located on it, where 0 is "no pain/bloating", 10 is "most severe pain/bloating you can imagine".
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mebeverine+Simethicone Combination | Mebeverine | Simethicone
Number analyzed (Participants) | 154 | 155 | 154
score on a scale | -3.65 (1.82) | -3.29 (1.91) | -3.11 (2.03)

4. Secondary Outcome: Change in Number of Days Per Week During Study Treatment Period When Drotaverine Was Taken.
Description: The data from last week of screening and run-in period was used for baseline assessment of number of days of drotaverin intake. Week 1, Week 2, Week3 and Week 4 assessments were the data from the last 7 days of the corresponding week.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Mebeverine+Simethicone Combination | Mebeverine | Simethicone
Number analyzed (Participants) | 152 | 154 | 152
number of days | -1.0 (2.3) | -1.1 (2.3) | -0.6 (2.3)

5. Secondary Outcome: Change in Quality of Life Evaluation Using IBSQOL Questionnaire Versus Baseline.
Description: Patients were asked to evaluate the quality of life using the Irritable bowel syndrome quality of life (IBSQOL) questionnaire at baseline at Visit 2 (Week 0) and at the end of the study treatment at Visit 3 (Week 4).
  The individual responses to the 34 items were summed and averaged for a total score and then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mebeverine+Simethicone Combination | Mebeverine | Simethicone
Number analyzed (Participants) | 154 | 155 | 154
score on a scale | -23.27 (21.19) | -19.57 (19.77) | -13.59 (16.83)

ADVERSE EVENTS:
Time Frame: Period for AEs collection was from the first study drug dose to the end of 30 days follow-up post-therapy period. Duration of treatment was 28 days.
Description: Any change to medical status, which occurred after study drug allocation at any dose in the specified study AE collection period were handled as an (S)AE. The post-therapy AE collection period was defined as 30 days after the subject's termination of study drug (collection of (S)AEs was passive in this period unless otherwise specified).
Arm/Group | Mebeverine+Simethicone Combination | Mebeverine | Simethicone
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/155 | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155 | 1/155 | 0/155
Other Adverse Events (participants affected / at risk) | 39/155 | 36/155 | 31/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mebeverine+Simethicone Combination (N=155) | Mebeverine (N=155) | Simethicone (N=155)
Covid-19 Pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mebeverine+Simethicone Combination (N=155) | Mebeverine (N=155) | Simethicone (N=155)
Headache (Nervous system disorders) | 23 | 18 | 20
Nausea (Gastrointestinal disorders) | 11 | 7 | 7
Asthenia (General disorders) | 5 | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT05175131/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT05175131/SAP_001.pdf